CLINICAL TRIAL: NCT07400757
Title: The Role of Statin and Vitamin D for the Treatment of Thyroid Eye Disease
Brief Title: Statin and Vitamin D Treatment in Patients With Thyroid Eye Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2025-08-018A
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Thyroid Eye Disease, TED; Graves Ophthalmopathy
Keywords: Thyroid Eye Disease; Graves Ophthalmopathy; Statin; Vitamin D; Atorvastatin; Autoimmune Disease; Inflammation; Randomized Controlled Trial; Factorial Design; Clinical Activity Score
MeSH Terms: conditions — Graves Ophthalmopathy; Autoimmune Diseases; Inflammation | interventions — Atorvastatin; Vitamin D

STUDY DESIGN:
Intervention Model Description: This study uses a 2×2 factorial, parallel-group design to evaluate the independent and combined effects of statin therapy and vitamin D supplementation. Participants are randomly assigned to one of four groups: standard care alone, statin plus standard care, vitamin D plus standard care, or combined statin and vitamin D plus standard care.
Masking Description: This is an open-label study. Neither the participants nor the investigators are blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care (No Intervention): Participants receive standard care for active thyroid eye disease according to current clinical practice for 24 weeks.
- Statin (Experimental): Participants receive standard care plus oral atorvastatin 20 mg once daily for 24 weeks.
  Interventions: Drug: Atorvastatin (Lipitor)
- Vitamin D (Experimental): Participants receive standard care plus oral vitamin D supplementation at a dose of 1400 IU daily for 24 weeks.
  Interventions: Dietary Supplement: Vitamin D
- Statin plus Vitamin D (Experimental): Participants receive standard care plus oral atorvastatin 20 mg once daily and oral vitamin D supplementation at a dose of 1400 IU daily for 24 weeks.
  Interventions: Drug: Atorvastatin (Lipitor); Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Atorvastatin (Lipitor) — Oral atorvastatin 20 mg administered once daily for 24 weeks.
  Arms: Statin; Statin plus Vitamin D
Dietary Supplement: Vitamin D — Oral vitamin D supplementation at a dose of 1400 IU administered once daily for 24 weeks.
  Arms: Statin plus Vitamin D; Vitamin D

SUMMARY:
The goal of this clinical trial is to learn whether statin therapy and vitamin D supplementation can improve disease activity in patients with active thyroid eye disease. The study will also evaluate the safety of these treatments. The main questions it aims to answer are:

* Does statin therapy reduce disease activity, as measured by changes in the Clinical Activity Score (CAS) and proptosis?
* Does vitamin D supplementation reduce disease activity in patients with active thyroid eye disease?
* Does combined treatment with statin and vitamin D provide greater improvement compared with either treatment alone or standard care?
* What side effects do participants experience during treatment?

Researchers will compare four groups: standard care alone, statin therapy plus standard care, vitamin D supplementation plus standard care, and combined statin and vitamin D therapy plus standard care.

Participants will:

* Be randomly assigned to one of four treatment groups
* Receive the assigned treatment for 24 weeks
* Attend clinic visits for clinical assessments and blood tests at baseline and at 24 weeks
* Be followed through medical record review for up to three years after completion of the intervention

DETAILED DESCRIPTION:
Thyroid eye disease (TED) is an autoimmune inflammatory disorder commonly associated with Graves' disease. The disease typically follows an active inflammatory phase, characterized by orbital inflammation, pain, redness, swelling, and progression of eye protrusion, followed by an inactive fibrotic phase with more permanent structural changes. Early intervention during the active phase is critical to reduce disease severity and prevent long-term functional and cosmetic complications.

Current treatments for active TED primarily focus on immunosuppression, such as systemic corticosteroids or other immunomodulatory therapies. However, these treatments may be associated with significant side effects and variable treatment responses. Therefore, there is an unmet need for adjunctive therapies with favorable safety profiles that may reduce disease activity and improve outcomes in patients with active TED.

Recent observational studies have suggested that statin use is associated with a lower risk of developing thyroid eye disease and a reduced severity of disease manifestations. These potential benefits appear to be independent of cholesterol-lowering effects and may be related to the anti-inflammatory and immunomodulatory properties of statins. In addition, vitamin D deficiency has been frequently observed in patients with TED, and vitamin D is known to play a role in immune regulation and inflammatory control. Experimental and clinical studies suggest that vitamin D supplementation may modulate autoimmune activity and reduce inflammatory responses.

Despite these findings, there is limited prospective clinical trial evidence evaluating the effects of statin therapy and vitamin D supplementation in patients with active TED. This study is designed as a randomized, open-label, 2×2 factorial clinical trial to evaluate the individual and combined effects of statin therapy and vitamin D supplementation on disease activity in patients with active TED.

Eligible participants with active TED will be randomly assigned to one of four groups: standard care alone, standard care plus statin therapy, standard care plus vitamin D supplementation, or standard care plus combined statin and vitamin D therapy. The intervention period will last for 24 weeks. Statin therapy consists of oral atorvastatin 20 mg once daily, and vitamin D supplementation consists of oral vitamin D at a daily dose of 1400 IU.

The primary outcomes of the study include changes in the Clinical Activity Score (CAS), improvement rate defined as a decrease of at least 2 points in CAS, changes in proptosis measured by Hertel exophthalmometry, and changes in thyroid-stimulating immunoglobulin (TSI) levels from baseline to 24 weeks. Secondary outcomes include changes in thyroid function, lipid profiles, blood glucose levels, and the use of thyroid-related medications and systemic corticosteroids during the intervention period.

Safety assessments will be conducted throughout the study by monitoring clinical symptoms, laboratory parameters, and reported adverse events. After completion of the 24-week intervention, participants will return to standard care and will be followed through medical record review for up to three years to observe long-term disease activity outcomes.

This study aims to provide prospective clinical evidence regarding the potential role of statin therapy and vitamin D supplementation as adjunctive treatments for active thyroid eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older
* Diagnosis of active thyroid eye disease with a Clinical Activity Score (CAS) of 3 or higher
* Low-density lipoprotein cholesterol (LDL-C) level of 100 mg/dL or higher

Exclusion Criteria:

* Prior orbital radiotherapy or orbital surgery for thyroid eye disease
* Use of statins or high-dose vitamin D supplementation (greater than 400 IU per day) within 3 months prior to enrollment
* Pregnancy
* Severe renal impairment, defined as an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73 m²

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Activity Score (CAS) | Baseline to 24 weeks
  Change in Clinical Activity Score (CAS)
Improvement Rate of Thyroid Eye Disease | Baseline to 24 weeks
  Proportion of participants achieving a decrease of ≥2 points in Clinical Activity Score (CAS)
Change in Proptosis | Baseline to 24 weeks
  Change in proptosis measured by Hertel exophthalmometry
Change in Thyroid-Stimulating Immunoglobulin (TSI) | Baseline to 24 weeks
  Change in serum thyroid-stimulating immunoglobulin (TSI) levels

SECONDARY OUTCOMES:
Change in Thyroid Function | Baseline to 24 weeks
  Change in thyroid function parameters (TSH, free T4, free T3)
Change in Lipid Profile | Baseline to 24 weeks
  Change in lipid parameters, including low-density lipoprotein cholesterol (LDL-C)
Change in Blood Glucose | Baseline to 24 weeks
  Change in blood glucose levels
Concomitant Medication Use | Up to 24 weeks
  Use of thyroid-related medications and systemic corticosteroids during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Sung Kuo, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data protection policies and ethical considerations related to participant privacy.

REFERENCES:
- [Background] Cardo C, Bernardo Santos R, Pinotti Pedro Miklos AB, Barbosa Jaconis S, Romaldini JH, Villagelin D. The relationship between cholesterol levels and thyroid eye disease. Eur Thyroid J. 2025 Feb 3;14(1):e240133. doi: 10.1530/ETJ-24-0133. Print 2025 Feb 1. PMID 39819487
- [Background] Chou YT, Lai CC, Li CY, Shen WC, Huang YT, Wu YL, Lin YH, Yang DC, Yang YC. Statin Use and the Risk of Graves' Orbitopathy: A Nationwide Population-Based Cohort Study. Thyroid. 2025 Feb;35(2):199-207. doi: 10.1089/thy.2024.0536. Epub 2025 Jan 13. PMID 39804287
- [Background] Wang CM, Chen YJ, Yang BC, Yang JW, Wang W, Zeng Y, Jiang J. Supplementation with active vitamin D3 ameliorates experimental autoimmune thyroiditis in mice by modulating the differentiation and functionality of intrathyroidal T-cell subsets. Front Immunol. 2025 Jan 30;16:1528707. doi: 10.3389/fimmu.2025.1528707. eCollection 2025. PMID 39949783